CLINICAL TRIAL: NCT06912750
Title: Effect of 4 7 8 Breathing Exercises With Teach Back Method on Pain Anxiety and Sleep Quality in Patients After Total Knee Arthroplasty: A Randomized Controlled Trial
Brief Title: 4-7-8 Breathing and Teach-Back Method for Pain, Anxiety, and Sleep After Knee Surgery: A Clinical Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erzurum Technical University (Other)
Responsible Party: Principal Investigator, Yasemin Erden, Assistant Professor, Erzurum Technical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 02.16.23.01.2025
Record Dates: First submitted 2025-02-25; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Patients With Total Knee Arthroplasty

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 4-7-8 Breathing Exercise with Teach-Back Method (Experimental)
  Interventions: Other: 4-7-8 Breathing Exercise with Teach-Back Method
- Standard Postoperative Care (No Intervention): In the control group, patients will complete the "Patient Information Form," the Visual Analog Scale (VAS) for pain, the State-Trait Anxiety Inventory (STAI), and the Richards-Campbell Sleep Questionnaire (RCSQ) before undergoing total knee arthroplasty, without any additional interventions beyond standard clinical protocols.
  Postoperatively, the VAS and STAI will be administered at the 6th, 12th, and 24th hours without any interventions. Following these assessments, patients will be asked to remain in a quiet and calm environment for 30 minutes. At the end of this period, the researcher will reassess pain and anxiety levels using the VAS and STAI, and the data will be collected. Additionally, at the 24th postoperative hour, the RCSQ will be administered, marking the conclusion of data collection for the control group.

INTERVENTIONS:
Other: 4-7-8 Breathing Exercise with Teach-Back Method — In the experimental group, patients will be provided with information regarding the purpose and significance of the 4-7-8 breathing technique using the Teach-Back method one day before surgery. To confirm comprehension, patients will be asked to repeat the information. The exercise will be demonstrated in a one-on-one session using the Teach-Back method, and patients will be guided through practical application. Following the training, patients will be instructed to perform the exercise independently, with the researcher monitoring its correct implementation. Each patient will be given a "4-7-8 Breathing Exercise Application Guide," which outlines the exercise steps based on relevant literature.
  Before surgery, patients will complete the "Patient Information Form," the Visual Analog Scale (VAS) for pain, the State-Trait Anxiety Inventory (STAI), and the Richards-Campbell Sleep Questionnaire (RCSQ). Postoperatively, the VAS and STAI will be administered both before (pre-test) and after
  Arms: 4-7-8 Breathing Exercise with Teach-Back Method

SUMMARY:
Total knee arthroplasty (TKA) is a surgical procedure performed to reduce pain and improve quality of life in elderly individuals with knee dysfunction due to osteoarthritis, rheumatoid arthritis, or other knee joint disorders. It is typically preferred in cases of advanced joint damage to help patients regain daily functional abilities. Postoperative rehabilitation is crucial for pain management, mobility, and overall recovery. The Teach-Back method is an effective educational technique that enhances patients' understanding of health information by encouraging them to repeat what they have learned. This approach improves information retention and promotes active participation in treatment, particularly among individuals with low health literacy. Complementary therapies, such as breathing exercises, can help manage common postoperative issues like pain, anxiety, and sleep disturbances. The 4-7-8 breathing technique has been shown to reduce anxiety and enhance sleep quality by regulating oxygen and carbon dioxide exchange. This method involves inhaling for four seconds, holding the breath for seven seconds, and exhaling for eight seconds, promoting physical and psychological relaxation.This study aims to evaluate the effects of 4-7-8 breathing exercises taught using the Teach-Back method on pain, anxiety, and sleep quality in patients undergoing total knee arthroplasty.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is a surgical intervention performed to alleviate pain and enhance quality of life in elderly individuals with impaired knee functionality due to osteoarthritis, rheumatoid arthritis, or other knee joint disorders. This procedure is primarily recommended in cases of advanced joint damage and aims to help patients regain their ability to perform daily activities. Postoperative rehabilitation plays a critical role in pain management, mobility improvement, and overall health recovery. The Teach-Back method is an effective educational strategy designed to enhance patients' comprehension of health-related information. This method ensures that patients accurately retain the information provided by healthcare professionals by requiring them to reiterate the learned content, thereby fostering active participation in their treatment process. Studies have demonstrated that this approach significantly improves information retention, particularly among individuals with low health literacy. Complementary therapies have been shown to be effective in managing common postoperative complications such as pain, anxiety, and sleep disturbances following TKA. Breathing exercises, in particular, have been found to reduce anxiety and improve sleep quality. Teaching breathing exercises through the Teach-Back method may contribute positively to the rehabilitation process by promoting both physical and psychological well-being. One such technique, the 4-7-8 breathing exercise, has been evidenced to aid in reducing anxiety and enhancing sleep quality. This technique involves inhaling for four seconds, holding the breath for seven seconds, and exhaling for eight seconds. By optimizing oxygen intake and facilitating the expulsion of carbon dioxide, this practice supports physiological and psychological relaxation. This study aims to evaluate the effects of 4-7-8 breathing exercises taught using the Teach-Back method on pain, anxiety, and sleep quality in patients undergoing total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are conscious and oriented,
* Able to communicate,
* Age 65 and over,
* No cognitive-mental problems,
* Standard Mini Mental Test (SMMT) score of 24 and above,
* Have not attended a course on breathing exercises and yoga before,
* Patients who agree to participate in the study verbally and in writing

Exclusion Criteria:

* Unconscious,
* Unable to communicate,
* Under 65 years of age

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Richard Campbell Sleep Quality Scale | 24 hours
  This scale evaluates the depth of night sleep, the time it takes to fall asleep, the frequency of waking up, the time it takes to stay awake when you wake up, the quality of sleep and the noise levels in the environment. When filling out the scale, the person is asked to mark the appropriate option for each item on a chart consisting of 6 items, each item being between 0 and 100. The scale is evaluated with the visual analog scale technique. The score between "0-25" from the scale indicates very bad sleep, and the score between "76-100" indicates very good sleep. The total score of the scale is evaluated based on the first 5 items. The 6th item evaluates the noise level in the environment and is not included in the total score evaluation. As a result, it is concluded that the sleep quality of the participants increases as the total score increases.
State Anxiety Scale | 24 hours
  The scale consists of 20 questions that measure state anxiety. The "State Anxiety Scale (STAI FORM TX-I, DKO)" requires the individual to express how he/she feels at a certain moment and under certain conditions. A minimum of 20 and a maximum of 80 points can be obtained from each subscale, with higher scores indicating a higher level of anxiety.
Visual Comparison Scale | 24 hours
  This scale, developed to determine the intensity of pain, is a 10 cm ruler scale with "No Pain" written on one end and "Unbearable Pain" on the other. It consists of numbers divided into equal intervals of one cm between the starting point where there is no pain and the point marked by the patient. In the evaluation of this scale, 0 = no pain, 1-4 = mild pain, 5-6 = moderate pain, 7-8 = severe pain and 10 = unbearable pain

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Erden, Assistant Professor, Study Director — Erzurum Technical University Faculty of Helath Science; Tülay Kılınç, Assistant Professor, Principal Investigator — Ataturk University Faculty of Nursing; Zeynep Bal, Principal Investigator — Firat University
Locations (1):
- Erzurum Techical University, Erzurum, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be openly shared. However, data may be available upon reasonable request and with appropriate ethical approval.